CLINICAL TRIAL: NCT00003708
Title: A Phase I Study of Cyclic Oral Administration of SCH 52365 for 21 of 28 Days in Patients With Advanced Solid Malignancies
Brief Title: Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Therapy and Research Center, Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066816; P30CA054174 (NIH); UTHSC-9785011336 (Other: UTHSCSA IRB); SACI-IDD-98-09 (Other: San Antonio Cancer Institute); SPRI-C98-247 (Other: Schering-Plough); NCI-V98-1502 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: temozolomide — Patients receive oral temozolomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated at escalating doses of temozolomide. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity (DLT) during courses 1 or 2, with at least 2 patients experiencing DLT at the next higher dose level.
  Other Names: Temodar; Temodal; Temcad

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of temozolomide in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, tolerability, maximum tolerated dose, and dose limiting toxicity of temozolomide in patients with advanced solid malignancies. II. Characterize the single- and multiple-dose pharmacokinetics of temozolomide following oral administration in these patients. III. Determine antitumor activity of temozolomide in these patients.

OUTLINE: This is an open label, dose escalation study. Patients receive oral temozolomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated at escalating doses of temozolomide. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity (DLT) during courses 1 or 2, with at least 2 patients experiencing DLT at the next higher dose level.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven solid malignancy for which no curative therapy exists Glioblastoma eligible if following criteria are met: Stable performance status Stable symptoms At least 4 weeks on stable dose of dexamethasone CNS metastases allowed if no progression or no new edema present Measurable or evaluable disease No acute or chronic leukemia or multiple myeloma No known bone marrow involvement with tumor

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT no greater than 3 times upper limit of normal (ULN) (5 times ULN if due to liver metastases) Renal: Creatinine no greater than 1.5 mg/dL Other: No malabsorption syndrome due to prior surgery, gastrointestinal disease, or other unknown reason No concurrent nonmalignant systemic disease No active uncontrolled infection No frequent vomiting or medical condition that could interfere with oral medication uptake (e.g., partial bowel obstruction, bowel resection, partial intestinal bypass, external biliary diversion) No prior or concurrent malignancies at other sites except carcinoma in situ of the cervix or adequately treated basal or squamous cell skin cancer HIV negative No AIDS-related illness Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No prior allogeneic, syngeneic, or autologous bone marrow transplantation No prior peripheral blood stem cell transplantation No concurrent biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered No concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy to at least 25% of bone marrow (including pelvic irradiation) and recovered No concurrent radiotherapy Surgery: Prior major gastrointestinal surgery allowed (e.g., Whipple procedure) Other: At least 4 weeks since any prior investigational therapy At least 24 hours since prior alcohol consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1998-07; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W. Tolcher, MD, Study Chair — San Antonio Cancer Institute
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas